CLINICAL TRIAL: NCT04308772
Title: Web-Based Physiotherapy Following Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/WS/0077
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Knee Arthroscopy; Physical Therapy
Keywords: knee; arthroscopy; physiotherapy; web-based

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Those randomised to the usual care arm will receive a leaflet which contains a standard programme of exercises Participants will be asked to complete their exercise programme as prescribed (at least once per day).
- Web-based physiotherapy (Experimental): Participants will receive a six week exercise programme, based on those in the usual care exercise sheet delivered via the web-based physio website (www.giraffehealth.com).
  Interventions: Behavioral: Web-based Physiotherapy

INTERVENTIONS:
Behavioral: Web-based Physiotherapy — Participants will receive an exercise programme, based on those patients usually get in the form of an exercise leaflet, delivered via a web-based physio website (www.giraffehealth.com). Participants will be asked to complete their exercise programme as prescribed (at least once each day) and to fill out an online exercise diary which the physiotherapist can see remotely from the clinical site.
  Arms: Web-based physiotherapy

SUMMARY:
Web-based physiotherapy might improve care following knee arthroscopy. For this study half of the participants will receive usual care (printed leaflet) and half will receive 6 weeks of web-based physiotherapy.

DETAILED DESCRIPTION:
Despite its minimally invasive nature, studies have shown that patients undergoing arthroscopic meniscectomy have pain, effusion, loss of range of motion, functional, neuromuscular and biomechanical changes, loss of quadriceps muscle strength, and a reduced quality of life (Durand et al.,1993;Goodwin and Morrissey,2003; Glatthorn et al.,2010). With changes in service delivery patients following arthroscopy only receive a printed leaflet. Web-based physiotherapy may offer offer cost effective support to patients. Therefore, the aim of this study is to undertake a single blind, randomised controlled pilot study examining the effectiveness of a six week web-based physiotherapy programme compared to usual care alone, for people following knee arthroscopy and to gather essential information for the planning of a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone Knee Arthroscopy surgery.
* Access to a personal computer/tablet or smart phone with an email address and internet connection
* Be able to understand English.

Exclusion Criteria:

* Infection or other post-operative complications
* Other significant co-morbidities for which exercise is contra-indicated
* Unwilling to be randomised to intervention/control group
* Taking part in another research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS). | Baseline to 6 weeks.
  The KOOS is a patient reported outcome measure, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It consists of 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).The KOOS is self-administered and takes approximately 10 minutes to complete. The KOOS is reliable, responsive to surgery and physical therapy and can be used to evaluate the course of knee injury and treatment outcomes (Roos et al.,1998).

SECONDARY OUTCOMES:
Change in Cincinnati Sports Activity Scale (CSAS) | Baseline to 6 weeks.
  CSAS is a patient reported outcome measure, developed to assess the patients' sports participation and identify patients who experience symptoms during athletic activities. It consists of 16 items in 5 separately scored subscales; the frequency of participation, the knee functions that occur during various sports activities and activities of daily living, the change that occurs in activity levels between treatment periods and the problems patients encounter with individual sports that place varying loads on the knee joint. The CSAS is self-reported and takes approximately 6 minutes to complete. The CSAS is reliable, valid and responsive and can be used to evaluate the sports activity levels and participation (Noyes et al., 1989).
Adherence to exercise programme | Weekly for 6 weeks
  Participants are advised to undertake their exercise programme at least once per day for six weeks and adherence will be based on the mean number of completed entries in exercise diaries over the 6 weeks of the programme and the total adherence to the programme will be calculated as a percentage.
Health Resource Form | Week 6
  a form detailing the number of interactions with health care professionals, such as physiotherapy and GP visits and medication use during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Nikologiannis, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No